CLINICAL TRIAL: NCT03923946
Title: STRICTLy CFT: A Feasibility Randomised Control Trial of a Compassion Focussed Therapy Intervention to Aid Recovery Post-stroke
Brief Title: STRICTLy CFT: a Compassion Focussed Therapy Intervention to Aid Recovery Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181002
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Stroke
Keywords: Stroke; Compassion Focused Therapy; CFT; Distress; Feasibility RCT
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Feasibility RCT
Masking Description: Due to the active nature of the interventions it is not possible to mask participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Compassionate Imagery Intervention- up to three 1:1 sessions, up to one hour each with the primary researcher
  Interventions: Behavioral: Compassion focused therapy
- Control (No Intervention): Treatment as usual arm

INTERVENTIONS:
Behavioral: Compassion focused therapy — Compassionate Imagery intervention based on compassionate imagery exercises in The Compassionate Mind Workbook by Irons and Beaumont, 2017
  Arms: Intervention

SUMMARY:
Individuals who have had a stroke are at greater risk of developing distress (e.g. depression and anxiety). These individuals are also likely to be highly critical of themselves as they are no longer able to do the things they used to be able to do.

Compassion Focused Therapy is a form of psychotherapy aimed at reducing an individual's self-criticism and increasing their self-compassion. CFT has been found to be effective at reducing distress in the general population and there is emerging evidence in the brain injury population. However, to date, there has not been a rigorous study to establish the effectiveness of CFT. Therefore, this feasibility randomised control trial aims to:

Establish the feasibility of recruitment, randomisation, and retention of participants; determine the acceptability and feasibility of a CFT intervention within a stroke population; determine the suitability of pre and post measures for assessing the impact of the intervention; Analyse the cost-effectiveness of the study; Establish effect sizes to enable an accurate estimation of the number of participants needed in a full scale RCT to find a treatment effect.

Individuals will be randomised into either a CFT intervention group, an active control arm (akin to a befriending type service) or a treatment as usual arm. Participants will receive up to three one hour sessions of CFT (intervention group) or befriending (active control group) or will not receive any additional support (treatment as usual group).

A total of 36 participants will be recruited, 12 in each arm of the study. Participants will be recruited from the Early Supported Stroke Discharge Teams within Derbyshire.

Participants will complete well-being, distress and self-criticism measures, pre, post and at 4 months follow-up. A semi-structured interview will also be conducted with a selection of participants from each arm.

DETAILED DESCRIPTION:
Stroke Stroke is a type of acquired brain injury (ABI) and is a heterogeneous term used to describe both ruptures to large blood vessels in the brain causing flooding with blood, and occlusions of tiny vessels in a part of the brain that is vital for functioning.

In the UK stroke is the second leading cause of death and disability, second only to coronary heart disease. Approximately 110, 000 strokes occur each year in England with prevalence rates estimated to be 7.20/1000.

Strokes can lead to changes in functioning in a variety of areas of life. As a result, individuals can often experience a range of emotional difficulties. For example, there is a high prevalence of mental health difficulties in stroke survivors; the most commonly reported are depression and anxiety disorders. Prevalence rates of distress vary between studies; however, it is estimated that the prevalence of post-stroke depression is approximately 31%, and post-stroke anxiety is estimated to be 18%. High levels of depression and anxiety can augment the functional impairments experienced as a result of a stroke. Depression in particularly is associated with reduced functioning outcomes and increased mortality rates.

In addition, studies have found high levels of self-criticism post-stroke as individuals realise they are no longer able to do things which they used to be able to. Studies have found higher rates of depression in individuals who continue to pursue what have now become unachievable life goals. It is postulated that this could be one of the reasons for the high prevalence rate of depression post-stroke, particularly if individuals do not re-evaluate their life goals to realign with any changes in cognitive capacity and functional deficits as a result of the stroke.

National Institute for Health and Care Excellence Guidance has suggested that individuals who have had a stroke should have access to psychological therapy to help with difficulties adjusting to life post-stroke. One such therapy is Compassion Focussed Therapy (CFT) which aims to reduce self-criticism by increasing self-compassion. CFT may be particularly effective in this population due to the specific challenges faced. For example, they have to adjust to the loss of previous functioning (both cognitively and otherwise) alongside managing the threat that a stroke may reoccur and the gradual and often frustrating nature of recovery which may be conditional on clinical input. The picture can then be complicated further by an individual's self-criticism tendencies which, as described above, can compound any challenges the individual is already facing. Therefore, CFT, which aims to reduce self-criticism and foster adjustment through self-compassion, would appear to be a well-suited intervention in this population.

CFT proposes a bio-psycho-social model of distress centred around three systems; a drive system, a threat system and a self-soothing system. The model suggests that an individual becomes distressed when the three systems become unbalanced. One of the ways this imbalance could happen is via self-criticism. Within this model, self-criticism is described as an internal threat and leads to an over-active threat-focused system. CFT focuses on reducing self-criticism by increasing the soothing system and reducing the threat system.

There is growing evidence to support this model of distress. For example, individuals in the general population who have high levels of self-criticism are also susceptible to developing mood related disorders like depression and anxiety.

Furthermore, high levels of self-criticism have been found to negatively impact on the effectiveness of psychological support unless self-criticism is specifically targeted.

There is also increasing evidence to support the effectiveness of CFT at reducing distress which will be discussed in further detail below.

There is a growing body of research which is showing promising results for CFT as an intervention for reducing distress in an ABI population.

There has been a collection of case studies conducted within this population utilising CFT to reduce symptoms of distress. Two of these studies found clinically meaningful reductions in distress scores post intervention. However, both of these studies utilised a CBT intervention in addition to CFT. Whilst reviews of the literature have found inconclusive evidence for the effectiveness of CBT alone to treat symptoms of distress in an ABI population, it is still unclear what direct impact the CFT intervention had. Nevertheless, Ashworth, (2015) found a reduction in symptoms that was approaching significance whilst utilising CFT alone.

O'Neill and McMillan (2012) utilised a single session compassionate imagery intervention in a group of individuals with an ABI. However, the authors failed to find a significant effect of single session compassionate imagery on empathy and self-compassion scores, although changes in self-compassion scores approached significance. It must be noted that this study only utilised a single session of compassionate imagery and did not assess the effect of this intervention on distress. Nonetheless, this study suggests compassionate imagery can be utilised in an ABI population and authors suggested future studies utilise repeated exposure to compassionate imagery to aid learning and retention.

Recently, researchers have conducted a naturalistic study with 12 individuals who received both group and individual CFT. This study found a significant reduction in depression and anxiety symptoms post CFT intervention which further suggests support for utilising CFT to reduce symptoms of anxiety and depression in an ABI population.

STUDY OBJECTIVES AND PURPOSE PURPOSE The aim of this study is to explore the feasibility of a full-scale trial to investigate the clinical and cost effectiveness of a compassion focussed intervention to manage distress post-stroke.

Whilst the research evidence in support of using CFT to reduce symptoms of distress post ABI is emerging, to date there has not been a Randomised Control Trial (RCT) conducted in an ABI or stroke population. The Medical Research Council (MRC) states there are certain stages that research needs to go through before conducting a definitive RCT, see Figure 2. Currently the research evidence meets the development stage. Therefore, feasibility/ pilot study is the next necessary step in the process.

There is evidence to suggest that the greatest risk of developing psychological distress is in the first few months post-stroke. This risk is then maintained throughout the first-year post-stroke and has a significant correlation to functional outcome. This review suggested that early diagnosis and treatment is therefore, vital for optimising recovery. Another more recent review found evidence that psychological interventions may prevent mood disorders post-stroke. Therefore, this study will explore CFT early on post-stroke.

PRIMARY OBJECTIVE The primary objective is to establish the feasibility of the study, including recruitment, randomisation, and retention of participants.

SECONDARY OBJECTIVE(S)

The secondary objectives are to:

* Determine the acceptability and feasibility of a compassionate imagery intervention within a stroke population.
* Determine the suitability of pre and post measures for assessing the impact of the intervention.
* Analyse the cost-effectiveness of the study.
* Establish effect sizes to enable an accurate estimation of the number of participants needed in a full scale RCT to find a treatment effect.
* Explore the effectiveness of the intervention OUTCOME MEASURES/ENDPOINTS PRIMARY OUTCOME MEASURE/ENDPOINT The primary outcome measures will be drop-out rates/ percentage completion rates and framework analysis from responses to interview questions about participants' experiences of being involved in the study.

SECONDARY ENDPOINTS/OUTCOMES The secondary outcome measures will include analysis of responses to psychometrics (including the HADS, WEWBS, EQ-5D, SCS) and service use questionnaires.

STUDY DESIGN A three-arm feasibility randomised control trial will be conducted comparing a compassion focussed intervention to an active control and usual stroke care. Participants will be randomised at baseline in equal proportions via a computer-generated programme developed to block randomise participants to an arm in the study.

Participants will be asked to complete standardised measures of distress (HADS), wellbeing (WEWBS), Quality of Life (EQ-5D) and self-compassion (SCS) at baseline, post-intervention and 4-month follow-up.

Participants will be invited to take part in a post-intervention interview; participants will be selected iteratively using purposive sampling to represent participants from all three arms and to include a range of severity of distress at baseline.

DATA ANALYSIS This study will utilise a mixed-methods approach for addressing feasibility objectives.

Quantitative data will be analysed using SPSS. Descriptive data will be analysed using Chi square and t-tests. Quantitative analyses will use a mixed linear model comparing distress, self-compassion and wellbeing scores at baseline versus 6-weeks and 4-month follow-ups, within and between the three allocation groups.

Interviews will be transcribed verbatim this may be completed by an outside company. If the post-intervention interviews are transcribed by a transcription service external to the University, a Transcriber Confidentiality Agreement will be completed with the chosen service. This will ensure that any of the information collected in the interviews will remain confidential. The chosen transcription service will be required to have a secure system for data transfer, access, and storage. Participants will be made aware that their interview will be sent for transcription at the consent stage of recruitment. If the interviews are not transcribed by an external company they will be transcribed by a member of the research team.

Interviews will be analysed using framework analysis (Ritchie & Spencer, 1994). Framework analysis allows both inductive and deductive analysis of the data.

STUDY SETTING Participants will be identified through NHS community stroke teams, hospital stroke wards and caseloads of community and acute stroke teams. Participants will be recruited from ESSD Teams within Derbyshire Community Healthcare Service NHS Foundation Trust and Derby Teaching Hospitals NHS Foundation Trust.

All participants will continue to receive their usual care alongside the study. The intervention arm will be delivered by the Primary Investigator and the active control arm will be delivered by volunteers from the local stroke association.

SELECTION OF PARTICIPANTS ELIGIBILITY CRITERIA Participants who have had a stroke will be invited to take part in the study after they have been discharged from the ESSD pathway.

Inclusion Criteria

Participants will be eligible for the study if they are:

• Eligible for the early supported discharge pathway this includes:

* Confirmed diagnosis of a new stroke.
* Over 18 Years old.
* Able to consent to being in the study.
* The patient and their family/carer agree to rehabilitation process continuing at home.
* The home environment is conducive to the community-based rehabilitation.
* Achievable rehabilitation goals can be identified.
* Document acknowledgement that the patient is sufficiently well enough from a medical perspective to be managed in the community.
* The patient's language and/or cognitive skills are at a level for them to manage on their own for periods as is necessary.

In addition to ESSD criteria participants must;

* Have a good grasp of the English language
* Have been discharged from the ESSD pathway Exclusion Criteria

Participants will be excluded if they:

* Have any communication difficulties that would prevent them from engaging in the intervention (including hearing impairments, visual impairments, inability to understand English). These will be assessed at researcher's discretion during baseline assessments.
* Had a diagnosis of dementia prior to the stroke.
* Are deemed to lack capacity to give informed consent. This will be judged via a qualified clinician.
* Have had previous experience of CFT
* Were receiving medical or psychological treatment for a mental illness at the time of their stroke.

Sampling This target sample-size should be feasible for the current study; the study will recruit from three ESSD teams in Derbyshire who each support up to 15 patients for 6 weeks. The Trust predicted that the ESSD teams would support 194 patients within the ESSD pathway per year. It is anticipated that all patients in the ESSD pathway will meet inclusion criteria for the study.

Size of sample Consistent with the feasibility-testing objectives of the study, sampling is based upon numbers required to estimate key design parameters. We will aim to recruit 12 participants per arm (36 participants in total), based on calculations demonstrating that these numbers would be sufficient to estimate relevant parameters with adequate precision (Julious, 2005).

Sampling technique Clinicians in the ESSD team will give all individuals they support information about the study and will pass the details those who show an interest on to the research team.

RECRUITMENT Potential participants for this study will be recruited via the Derbyshire NHS Stroke Services. Participants will be recruited over a 13-month time-period.

Participants will be approached by clinicians within Derbyshire NHS Stroke Services about the study. Clinicians will provide potential participants with information about the study and pass on the contact details of those who express an interest in participating to the research team. The research team will then arrange a suitable time to either meet with the participant or have a phone conversation to talk through the study and ensure they understand what will be required of them.

It will be explained to the potential participant that entry into the trial is entirely voluntary and that their treatment and care will not be affected by their decision. It will also be explained that they can withdraw at any time, but attempts will be made to avoid this occurrence. In the event of their withdrawal it will be explained that their data collected so far may not be erased in accordance with the University's Research Privacy Notice and information given in the Participant Information Sheet and we will seek consent to use the data in the final analyses where appropriate.

RANDOMISATION AND BLINDING Participants will be randomised at baseline (after informed consent and baseline assessments) in equal proportions to the CFT intervention, active control, or usual stroke care once the individual has consented to taking part in the study. A computer-generated programme will be developed to block randomise participants to an arm in the study. This will be done via an allocation sequence and an email will be sent to the researcher to inform them which arm the participant is in.

It is not pragmatically possible for the participant or therapist to be blinded to group allocation due to the active nature of the intervention.

STUDY REGIMEN Individuals will complete baseline measures before being randomly allocated to one of three arms. These will either be completed online, face to face, over the phone or via postal forms, depending on participant preference and communication needs.

Once an individual has been randomly allocated to a treatment arm the researcher will contact them via a phone call to inform them which arm they have been allocated to. A follow-up letter will be sent to aid recall. If a participant withdraws from the study after they find out which arm they have been allocated they will not be replaced in the study as acceptability of randomisation is one of the outcomes of interest in this feasibility study.

Researchers will also conduct post-intervention interviews at four-months and post-measures at six-week and four-month follow up.

Participants in each arm will also receive care as usual based on the discharge report from the ESSD team from the neurological outpatient therapy service.

Intervention arm- compassionate imagery Based on previous literature, namely O'Neill and McMillan (2012), the compassion focussed intervention will be based on compassionate imagery. As suggested by the researchers in this study, the intervention will be delivered over a number of sessions to aid learning and retention.

A researcher will meet with the individual for up to three sessions and deliver a compassionate imagery intervention. The first session will be face to face with the option of delivering the other two sessions remotely (either via Skype or phone calls). It is important to conduct the first session face to face so that the intervention can be adapted as needed depending on the ability/needs of the participant. The other two sessions may be delivered remotely depending on the researcher's time constraints and participant preference.

Participants will be asked if they would like to take a copy of the recording or script home with them after the first session to practice. This will allow the researcher to troubleshoot any potential problems during the second and third sessions. The participant will keep the script/ recording for the duration of the study and will have the option to keep this after the study is completed.

During the intervention, the participant will be asked to create a compassionate image. Compassionate imagery works on the premise that we can stimulate different systems in our brain by imagining certain situations/ pictures. For example, if you are hungry and imagine a nice meal, you will activate the same bodily systems as if the meal were right in front of you. The same premise works for imagining threatening stimuli; our own self-talk and images we create in our head can lead to an activation in the threat system. The same can be said for compassion; if we imagine someone saying kind and reassuring words to us, it can activate the soothing system within our brain. Compassionate imagery therefore, encourages an individual to be self-compassionate and kinder to ones-self in order to reduce the threat system (see Gilbert, 2010 for further description).

The participant will be asked to create a compassionate other/ place that is wise, warm, strong and non-judgemental. Someone or something that wants the best for you, provides unconditional love and gives encouragement. The aim of this is to stimulate the self-soothing system and to reduce self-criticism. See Intervention script 181002 for the proposed intervention script for this study.

It is postulated that three sessions will be an effective way to deliver the intervention based on clinical judgment of psychologists working within the Derbyshire NHS stroke team.

Researchers will not place restrictions on carers being present during the intervention sessions. However, the researcher will monitor the carer's influence on the session and reserves the right to ask the carer to leave if they are adversely affecting the intervention.

Service-user involvement; Researchers have held a consultation meeting with a stakeholder group: to ascertain the feasibility of delivering this intervention and to highlight any barriers they envisage. The proposed intervention has been refined accordingly.

Active control arm The details of participant's who have been consented in to the study and randomised to the control arm will be passed on to volunteers from a local stroke association group who have agreed to provide a befriending service. These volunteers have a good working relationship with the Derbyshire NHS Trust and have up to date DBS checks to meet with patients in their own homes. Volunteers have also attended training programmes as part of the work they currently do with Derbyshire NHS Trust. The volunteer will then contact participants to arrange to either meet that participants in a place that is convenient for them or have a phone conversation at a convenient time for them. If the participant decided it is more convenient to meet outside of their home, travel and parking expenses will be paid for the participant and volunteer by the research team.

Participants will meet or talk to the volunteer for up to three sessions. These will occur once a week for up-to one hour-per-week and will be recorded for content via a Dictaphone. Participants will receive befriending support from the same volunteer throughout the study.

Carers will be asked not to be present for these sessions to reduce burden on the volunteers.

It is envisaged that participants and volunteers will discuss themes around recovery, loss of self and role, and re-gaining valued roles.

Treatment as usual arm Participants will be contacted by the researcher to inform them that they have been allocated to the treatment as usual arm and reminded what this entails. They will also be reminded that they will be contacted again in six weeks and four months to completed post measures.

Post intervention interviews Qualitative interviews will be conducted with 6-8 participants (3-4 per arm) to provide a description of the acceptability of the design and procedures of the trial (see Interview script 181002 for interview scripts).

Informed consent for interviews will be obtained at the start of the study. Participants will be selected iteratively using purposive sampling to represent participants from all three arms and to include a range of severity of distress at baseline. Interviews will be recorded, and consent confirmed at the start of the interview. Interviews will be conducted by an external researcher and transcribed by the lead researcher.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for the early supported discharge pathway this includes:

  * Confirmed diagnosis of a new stroke.
  * Over 18 Years old.
  * Able to consent to being in the study.
  * The patient and their family/carer agree to rehabilitation process continuing at home.
  * The home environment is conducive to the community-based rehabilitation.
  * Achievable rehabilitation goals can be identified.
  * Document acknowledgement that the patient is sufficiently well enough from a medical perspective to be managed in the community.
  * The patient's language and/or cognitive skills are at a level for them to manage on their own for periods as is necessary.

In addition to ESSD criteria participants must;

* Have a good grasp of the English language
* Have been discharged from the ESSD pathway

Exclusion Criteria:

* Participants will be excluded if they:

  * Have any communication difficulties that would prevent them from engaging in the intervention (including hearing impairments, visual impairments, inability to understand English). These will be assessed at researcher's discretion during baseline assessments.
  * Had a diagnosis of dementia prior to the stroke.
  * Are deemed to lack capacity to give informed consent. This will be judged via a qualified clinician.
  * Have had previous experience of CFT
  * Were receiving medical or psychological treatment for a mental illness at the time of their stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of an RCT design | 4 months (per participant)
  Answers from post-intervention interviews

SECONDARY OUTCOMES:
distress | 6 weeks
  Analysing pre-post scores on the Hospital Anxiety and Depression Scale (HADS). The HADS has two sub-scales; an anxiety sub-scale and a depression sub-scale (both range from 0-21, with higher scores indicating more distress).
well-being | 6 weeks
  Analysing pre-post scores on the Warwick Edinburgh Mental Well-being Scale (WEMWBS). A total score is calculated by summing answers on all questions and ranges form 14-70 with higher scores indicating greater well-being.
Process | 6 weeks
  Analysing pre-post scores on the Self-Compassion Scale (SCS). This scale has 4 sub-scales. Subscale scores are computed by calculating the mean of subscale item responses. To compute a total self-compassion score, reverse score the negative subscale items before calculating subscale means - self-judgment, isolation, and over-identification (i.e., 1 = 5, 2 = 4, 3 = 3. 4 = 2, 5 = 1) - then compute a grand mean of all six subscale means. Researchers can choose to analyze their data either by using individual sub-scale sores or by using a total score. Subscale scores range form 5-25 with higher scores indicating more compassion.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Derbyshire Community Hospitals, Derby
  - Royal Derby Hospital, Derby

IPD SHARING:
Plan to Share IPD: No